CLINICAL TRIAL: NCT02698423
Title: Human Papillomavirus Testing Versus Liquid-based Cytology for Non-attendees of Cervical Cancer Screening: Results of a Randomised Controlled Trial
Brief Title: Feasibility and Acceptability of Offering Self-sampling to Non-attendees in Primary Care
Acronym: DEPIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Prof. Patrick Petignat, Professor, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CER 11-034
Record Dates: First submitted 2016-02-23; First posted 2016-03-03 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Cancer of the Uterine Cervix
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cobas HPV DNA test (Experimental): Women will be invited to perform HPV self-testing with the Cobas HPV DNA test at home.
  Interventions: Device: Cobas HPV DNA Test
- Papanicolau test (Active Comparator): Women will be invited to come to the hospital to undergo a Papanicolau test (Pap test), which will be performed by the clinician.
  Interventions: Other: Papanicolau test

INTERVENTIONS:
Device: Cobas HPV DNA Test — Women will receive a home-sent sample for HPV self-testing
  Arms: Cobas HPV DNA test
Other: Papanicolau test — Women will be invited to come in for a physician-performed Pap test
  Arms: Papanicolau test

SUMMARY:
The purpose of this study is to determine whether human-papillomavirus (HPV) self-sampling can be used as a primary screening test for unscreened women.

DETAILED DESCRIPTION:
Women residing in the canton of Geneva, aged between 25 and 69 years, who haven't had a Pap test in the last three years, will be invited to participate. Participation to the study will be encouraged through public displays, social networks, and medical consultations. Women meeting the eligibility criteria will be enrolled in the study. They will be randomized into two groups and will receive a home-sent letter, inviting them to either come in for a Pap test or to perform and send back the HPV self-sample that they'll receive at their domicile. Both groups will also receive a questionnaire, in order to better understand the reasons for their previous non-attendance to cervical cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* No previous cervical cancer screening test in the last three years

Exclusion Criteria:

* pregnancy
* previous hysterectomy

Ages: 25 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2011-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
Data will be used for scientific publications.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cobas HPV DNA Test | Papanicolau Test
Started | 336 | 331
Completed | 317 | 307
Not Completed | 19 | 24
Not completed — Lost to Follow-up | 19 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cobas HPV DNA Test | Papanicolau Test | Total
Number analyzed (Participants) | 336 | 331 | 667
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (10.9) | 42.1 (10.8) | 42.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 336 | 331 | 667
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 105 | 106 | 211
  Not Hispanic or Latino | 231 | 225 | 456
  Unknown or Not Reported | 0 | 0 | 0
Relationship Status [Count of Participants; unit: Participants]
  With a partner | 161 | 154 | 315
  Single | 175 | 177 | 352

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Performed HPV Self-testing Compared to the Number of Participants Who Responded to the Invitation to Come to the Hospital for Pap Testing
Description: Compare the participation rate to cervical cancer screening for home-based human papillomavirus testing based on self-sampling versus clinic-based, physician-performed Pap testing.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Cobas HPV DNA Test: Women will be invited to perform HPV self-testing with the Cobas HPV DNA test at home.
  Cobas HPV DNA Test: Women will receive a home-sent sample for HPV self-testing. N=336
- Papanicolau Test: Women will be invited to come to the hospital to undergo a Papanicolau test (Pap test), which will be performed by the clinician.
  Papanicolau test: Women will be invited to come in for a physician-performed Pap test.
  N=331
Arm/Group | Cobas HPV DNA Test | Papanicolau Test
Number analyzed (Participants) | 336 | 331
Participants | 317 | 307

2. Secondary Outcome: Proportion of Women With a Positive HPV Self-test Who Underwent All the Recommended Follow-up Clinical Investigations.
Description: Assess the compliance with further follow-up among women having tested positive for the presence of HPV at baseline screening.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cobas HPV DNA Test | Papanicolau Test
Number analyzed (Participants) | 336 | 331
Participants | 317 | 307

ADVERSE EVENTS:
Description: Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Arm/Group | Cobas HPV DNA Test | Papanicolau Test
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes